CLINICAL TRIAL: NCT05914467
Title: A Randomized Trial Investigating the Superiority of TDM-optimized Teicoplanin Dosing Versus Standard of Care
Brief Title: TDM-optimized Teicoplanin Dosing Versus Standard of Care
Acronym: PLATO-3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113998; 2023-503411-15-00 (Other: EU CT-number)
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Teicoplanin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 between standard treatment and treatment guided by TDM with MIPD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Participants receive teicoplanin on discretion of the doctor
- Model Informed Precision Dosing (MIPD) guided Therapeutic Drug Monitoring(TDM) (Experimental): Participants start on standard of care dosing. After 2 days blood samples will be analysed and exposure will be determined using MIPD. Wherever necessary dose adjustments will be made.
  Interventions: Drug: Teicoplanin

INTERVENTIONS:
Drug: Teicoplanin — Dose will be adjusted in the study arm using MIPD guided TDM- dosing
  Arms: Model Informed Precision Dosing (MIPD) guided Therapeutic Drug Monitoring(TDM)

SUMMARY:
Value of TDM for teicoplanin is not well defined. In this single-center low-interventional randomized trial the investigators aim to investigate the superiority of teicoplanin TDM-optimized using Model-Informed-Precision-Dosing (MIPD) of unbound concentrations versus the standard of care (dosing based on antibiotic guidelines) in target attainment.

DETAILED DESCRIPTION:
Teicoplanin is a glycopeptide antibiotic that is frequently used in the treatment of gram-positive bacterial infections.

The glycopeptide antibiotic vancomycin is currently the first choice of treatment against methicillin-resistant Staphylococcus aureus (MRSA), but teicoplanin is found to have a similar efficacy while showing less nephrotoxicity (4.8% vs 10.7%). Vancomycin dosing is based on therapeutic drug monitoring (TDM). In contrast to vancomycin, value of TDM for teicoplanin is not as well defined. In this study the superiority of teicoplanin TDM-optimized dosing using Model-Informed-Precision-Dosing (MIPD) of unbound concentrations versus the standard of care (dosing based on antibiotic guidelines) in target attainment will be investigated. The overall aim of this research is to improve antibiotic treatment with teicoplanin to allow safe and optimal treatment of glycopeptide susceptible strains and to prevent de novo development of resistance.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is admitted to the ICU, haematology, gastroenterology or orthopaedics department.
2. The patient is at least 18 years old on the day of inclusion.
3. The patient is treated with teicoplanin as part of standard care.
4. The patient or a representative is willing to sign the Informed Consent Form

Exclusion Criteria:

1. The patient has previously participated in this study.
2. The patient receives any form of renal replacement criteria (RRT) other than CVVHD / CVVHDF.
3. Expected duration of teicoplanin therapy is less than 5 days.
4. The patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Fraction of participants that reaches therapeutic exposure after 5 days of treatment | 5-7 days after initiation of teicoplanin therapy
  Unbound teicoplanin exposure after 5 days will be determined and compared to the predefined therapeutic window of 70-150 mg/L*24h

SECONDARY OUTCOMES:
Time until reaching target attainment | 5-7 days after initiation of teicoplanin therapy
  Time until a participant reaches the therapeutic window will be estimated using the MIPD
Clinical failure | 30 days after initiation of teicoplanin therapy
  Incidence of clinical failure at day 30. Incidence of clinical failure of teicoplanin treatment will be defined as occurrence of one of the following on day 30:
  * Persistent bacteremia
  * Uncontrolled infection at the site of infection by the pathogen for which teicoplanin treatment was started
  * Escalation of therapy
  * Switch of antimicrobial therapy due to lack of effectiveness of teicoplanin
Days in hospital | 30 days after initiation of teicoplanin therapy
  Total number of days in the hospital

OTHER OUTCOMES:
Acute Kidney Injury (AKI) | 30 days after initiation of teicoplanin therapy
  incidence of AKI during teicoplanin treatment. Occurrence of nephrotoxicity will be defined as a binary denominator complying to any of the following markers according to the Kidney Disease: Improving Global Outcomes (KDIGO) guideline for acute kidney injury.
  * Increase in serum creatinine of > 0.3 mg/dl within 48 hours
  * Increase in serum creatinine to > 1.5 times baseline, which is known or presumed to have occurred within the prior 7 day

CONTACTS AND LOCATIONS:
Overall Officials: Nynke Jager, Principal Investigator — Radboud university medical center (Radboudumc)
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No